CLINICAL TRIAL: NCT04734704
Title: Defining the Role of the Skin Microbiome in Vitiligo and Immune-related Adverse Events in Advanced Melanoma Patients Treated With Anti-PD1
Brief Title: Defining the Role of the Skin Microbiome in Immune-related Adverse Events
Acronym: SKINBIOTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/41
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Vitiligo; Skin Melanoma
Keywords: immunotherapy; checkpoint inhibitors; vitiligo; skin microbiota; metastatic melanoma.
MeSH Terms: conditions — Vitiligo; Melanoma

STUDY DESIGN:
Intervention Model Description: Prospective, Monocentric (CHU de Bordeaux, Department of dermatology ), with 4 groups :
  * vitiligo patients
  * Metastatic melanoma patients receiving anti-PD-1 but without cutaneous irAEs
  * Metastatic melanoma patients receiving anti-PD-1 who developed vitiligo lesions
  * metastatic melanoma patients who developed vitiligo under anti-PD-1, who discontinued the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- vitiligo patients (Experimental): Adult patients diagnosed with Vitiligo according to usual criteria
  Interventions: Procedure: skin swabs at lesional and non-lesional sites
- metastatic melanoma patients under anti-PD-1 who did not develop cutaneous irAEs (Experimental): metastatic melanoma patients under anti-PD-1 who did not develop Cutaneous Immune-Related Adverse Events (cutaneous irAEs).
  Interventions: Procedure: skin swabs on skin
- Metastatic melanoma patients under anti-PD-1 who developed vitiligo lesions (Experimental): patients with metastatic melanoma, under anti-PD-1 who developed vitiligo lesions
  Interventions: Procedure: skin swabs at lesional and non-lesional sites
- metastatic melanoma patients with vitiligo lesions under anti-PD-1 who discontinued (Experimental): Metastatic melanoma who developed vitiligo lesions under anti-PD-1 who discontinued the treatment
  Interventions: Procedure: skin swabs at lesional and non-lesional sites

INTERVENTIONS:
Procedure: skin swabs at lesional and non-lesional sites — It will be examined in patients skin swabs sampled at lesional and non-lesional sites
  Arms: Metastatic melanoma patients under anti-PD-1 who developed vitiligo lesions; metastatic melanoma patients with vitiligo lesions under anti-PD-1 who discontinued; vitiligo patients
Procedure: skin swabs on skin — It will be examined in patients skin swabs sampled on skin
  Arms: metastatic melanoma patients under anti-PD-1 who did not develop cutaneous irAEs

SUMMARY:
The skin microbiome has been implicated in several cutaneous autoimmune pathologies such as psoriasis and atopic dermatitis. However, its role in vitiligo and vitiligo lesions occuring in patients receiving anti-PD-1 for metastatic melanoma

DETAILED DESCRIPTION:
Melanoma is the most dangerous skin cancer accounting for the highest skin cancer deaths. The prognosis for metastatic melanoma has improved considerably in recent years thanks to advances in the field of immunotherapy. The development of molecules blocking certain immunological "checkpoints" (checkpoints exerted by the CTLA-4 (Cytotoxic T lymphocytes Associated protein 4) and PD-1 (Programmed cell Death protein 1) has made it possible to obtain a significant improvement of the overall survival (OS) of patients treated for metastatic melanoma. Ipilimumab, an antibody blocking CTLA-4, is the first immunotherapy marketed, demonstrating for the first time a therapeutic response, however in a small number of patients (10 to 15%) and with significant toxicity (25% of grade 3-4). Subsequently, a second generation of more effective checkpoint blockers (30 to 40% good response) and less toxic, anti-PD-1 antibodies (pembrolizumab and nivolumab), quickly obtained a marketing authorization in the first line treatment of metastatic melanoma treatment and recently in an adjuvant situation after lymph node dissection in order to limit the risk of recurrence. However, despite these advances, a certain number of patients do not respond to treatment and it remains difficult to predict this therapeutic response. Furthermore, patients treated with ICI often experience cutaneous immune-related adverse events manifesting as skin rash, dermatitis, epidermal necrolysis, and in some cases as vitiligo like depigmentation of the skin, testifying to the development of a specific immunogenicity towards the melanocytes, cells causing melanoma, and responsible for a discoloration of the skin. Several studies have reported that a modification of certain bacteria in the digestive microbiota was predictive of the antitumor response to immunotherapy, while others were predictive of the appearance of significant autoimmune ICI-related toxicities (colitis). Several phase 1 studies have evaluated the impact of taking probiotics or fecal transplants on the tumor response of patients receiving immunotherapy for cancer (NCT 03819296; NCT03817125; NCT03643289). Thus by these new concepts, it would be interesting to assess the composition of the skin microbiota in patients treated with anti-PD-1 immunotherapy for the management of metastatic melanoma and developing during their follow-up vitiligo; predictive side effect of improved survival. These data will be compared to those obtained from patients with common vitiligo. This will be examined in patients skin swabs sampled at lesional and non-lesional sites. Functionally, we will characterize the microbial pathways using shotgun sequencing of microbial genomes and meta-transcriptomics (RNA sequencing of microbial communities of the skin).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with Vitiligo according to usual criteria.
* Adult patients with metastatic melanoma, under anti-PD-1 who developed vitiligo
* Adult patients with metastatic melanoma who did not develop Immune related adverse events under anti-PD-1
* Adult patients with metastatic melanoma who developed vitiligo under anti-PD-1 and discontinued the treatment
* Free, informed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patients under 18 years old.
* No treatment for vitiligo in the past 4 weeks
* Patients under legal protection or unable to express their consent.
* Patients not affiliated to a health insurance system.
* Patients deprived of liberty by judiciary or administrative decision or hospitalized without consent or admitted in a sanitary or social institution for another reason than research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Determine skin microbiota by sequencing with vitiligo in advanced melanoma patients under immune-checkpoint inhibitors (ICI) immunotherapy. | Day 1
  The composition of the skin microbiota will be characterized on skin swabs using shotgun sequencing of microbial genomes and meta-transcriptomics (RNA sequencing of microbial communities of the skin).

CONTACTS AND LOCATIONS:
Overall Officials: Julien SENESCHAL, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Dermatologie - Hôpital Saint-André, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No